CLINICAL TRIAL: NCT04550910
Title: Randomized Clinical Trial Comparing Two Adjuvant Radiotherapy Hypo Fractionation Schedules In The Treatment of Post Mastectomy Breast Cancer Patients
Brief Title: RCT Comparing 2 Radiotherapy HypoFractionation Schedules In Breast Cancer Patients
Acronym: Breastcancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Momen Elsayed Hassan, MSc., Assistant Lecturer of Radiation Oncology, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RO1912-30902
Record Dates: First submitted 2020-08-18; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Radiotherapy Side Effect; Locoregional Recurrence
Keywords: Post Op radiotherapy; Mastectomy; Locoregional Control
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): 40 Gy /15 fx / 3 weeks, 5 days per week, is a dose prescribed (after randomization ) for Breast Cancer patients indicated for adjuvant RTH after mastectomy
  Interventions: Radiation: Hypofractionation Schedules for Breast Cancer patients after mastecomy
- Arm B (Experimental): 28.5 Gy delivered in 5 once-weekly fractions of 5.7 Gy is a dose prescribed (after randomization )for Breast Cancer patients indicated for adjuvant RTH after mastectomy
  Interventions: Radiation: Hypofractionation Schedules for Breast Cancer patients after mastecomy

INTERVENTIONS:
Radiation: Hypofractionation Schedules for Breast Cancer patients after mastecomy — Two Radiotherapy HypoFractionation Schedules will be applied, after randomization, for female breast cancer patients after mastectomy.

SUMMARY:
This is a prospective randomized Phase III trial to assess efficiency of two post mastectomy hypofractionation schedules (40 Gy /15 fx / 3 weeks, 5 days per week VS 28.5 Gy delivered in 5 once-weekly fractions of 5.7 Gy each week) as adjuvant radiotherapy in female patients with breast cancer after mastectomy.

DETAILED DESCRIPTION:
166 patients of breast cancer patients after mastectomy ( 83 patients in each arm ) will be randomize into 2 hypofractionation arms : Arm A: 40 Gy /15 fx / 3 weeks, 5 days per week . Arm B: 28.5 Gy delivered in 5 once-weekly fractions of 5.7 Gy each week.

Simulation:

Patient will be simulated on CT simulator using breast wedge with angle. Serials will be taken every 2 mm from upper neck down to mid abdomen.

Contouring:

CTVcw, CTVRNI will be contoured through RTOG guidelines . PTV is added as 0.5 cm all around CTV. Lungs, Heart, brachial plexus, spinal cord, esophageus and thyroid will be contoured as OAR. (www.rtog.org/CoreLab/ContouringAtlases/BreastCancerAtlas.aspx).

D)Dose Constraints:

Arm A:

PTV EVAL ( CW) : V90 % ≥ 90 %. - V105 % ≤ 5% - V107%≤ 3 %. Ipsilateral lung: V20 less than 20-25% - V 8 less than 35%- Contra lateral lung: V4 less 10 %. Heart: V16 less than 5% (Lt sided). V20 less than 5% (Lt sided). V16 is 0%.(Rt sided) V20 is 0% (Rt sided). Mean heart dose ≤ 320-400 cGy. Contra lateral breast : D max≤ 240 cGy. V 144 cGy less than 5 %. SCV : V90 % ≥ 90 %. Thyroid : Mean dose less than 35 Gy - V30 less than 50 %.

Arm B:

PTV EVAL ( CW) : V90 %≥ 90 %. - V105 %≤ 5% - V107%≤ 2 %.

Ipsilateral lung: V30%less than 15 -20% - V15% less than 30-35% - V5 % less than 50-55%.

Contra lateral lung : V5 % less than 5%. Heart :V25 % less than 5 % - V5 % less than 30 - 35 %. Contra lateral breast: V3 % less than 5 %. SCV : V90 % ≥ 90 %.

Follow up:

A)Weekly follow up will be done during sessions then regular clinical exam every 3 months to assess :

1. Acute and late toxicity regarding pain, pulmonary toxicity, dysphagia, skin toxicity and lymphedema.Assessment will be done according to RTOG and CTCv.5.
2. Any local (chest wall) recurrence, regional (nodal) recurrence.

B)Annual Mammogram. C)Any another investigation (once indicated)

ELIGIBILITY:
Inclusion Criteria:

* Invasive carcinoma of the breast.
* Complete microscopic excision of primary tumour and axillary dissection or SLNB .
* Females with locally advanced breast cancer ( T3/T4 or N + or both ) who are candidate for neoadjvant chemotherapy regardless pathological stage after mastectomy.
* Patients with pathological stage (T3/ T4, +/- N+) or ( N+, any T) after upfront mastectomy.
* Able to comply with follow up.
* Written informed consent

Exclusion Criteria:

* Patients do not match with inclusion criteria.
* Collagen vascular disease, specifically systemic lupus, or scleroderma.
* Pregnancy or lactation at the time of radiotherapy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Chest wall pain | 3 months form starting of Adjuvant radiotherapy to chest wall.
  Grades of toxicity will be assessed according to The Radiation Therapy Oncology Group (RTOG) morbidity scoring criteria. Scoring starts with low grade toxicity sacle ( Grade 1 or 2) while Grade 3 or 4 considered High grade toxicity.
Dysphagia | 3 months form starting Adj radiotherapy to chest wall.
  Grades of toxicity will be assessed according to The Radiation Therapy Oncology Group (RTOG) morbidity scoring criteria. Scoring starts with low grade toxicity sacle ( Grade 1 or 2) while Grade 3 or 4 considered High grade toxicity.
Skin | 3 months form staring adjvant radiotherapy to chest wal.
  Grades of toxicity will be assessed according to The Radiation Therapy Oncology Group (RTOG) morbidity scoring criteria. Scoring starts with low grade toxicity sacle ( Grade 1 or 2) while Grade 3 or 4 considered High grade toxicity.
Pulmonary Toxicity | Assessment will be started 6 months after end of adjuvant radiotherapy to chest wall then Biannaully for 2 years.
  Grades of toxicity will be assessed according to The Radiation Therapy Oncology Group (RTOG) morbidity scoring criteria. Scoring starts with low grade toxicity sacle ( Grade 1 or 2) while Grade 3 or 4 considered High grade toxicity.
Brachial plexopathy | Assessment will be started 6 months after end of adjuvant radiotherapy to chest wall then Biannaully for 2 years.
  Grades of toxicity will be assessed according to The Radiation Therapy Oncology Group (RTOG) morbidity scoring criteria. Scoring starts with low grade toxicity sacle ( Grade 1 or 2) while Grade 3 or 4 considered High grade toxicity.
Lymphedema | Assessment will be started 6 montha form ending adjuvant radiotherapy to chest wall and axilla then then Biannaully for 2 years.
  Common Toxicity Criteria v.5 ( Arm volume at CC.Grading done according to Interlimb Volume Difference.Interlimb volume difference > 30 % is considered Grade 3 Lymphedema) and Cheng scale ( To detect proportion of patients having moderate or severe lymphedema (Grade 》II)

SECONDARY OUTCOMES:
Local control | Annually after the end of chest wall irradiation for 2 years. ] must be confirmed by cytological/ histological assessment
  Local Recurrence Rate (LCR) including ipsilateral chest wall +/- regional nodal recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Osama Yousof, MD, Principal Investigator — National Cancer Institute, Egypt
Locations (1):
- NCIEGYPT, Cairo, Fom Elkhalig, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: First results of the randomised UK FAST Trial of radiotherapy hypofractionation for treatment of early breast cancer (CRUKE/04/015): The FAST Trial lists group. Radiotherapy and Oncology, 100(1), pp.93 — http://www.thegreenjournal.com/article/S0167-8140(11)00337-9/pdf
- See also: FAST Trial Finds Long-Term Side Effects Similar for Once-Weekly and Conventional Breast Radiation Therapies — http://www.ascopost.com/News/59403